CLINICAL TRIAL: NCT06773013
Title: Safety and Effectiveness of Sonu Acoustic Resonance Therapy for the Treatment of Pediatric Patients With Moderate to Severe Nasal Congestion.
Brief Title: Safety and Effectiveness of Sonu for Pediatric Nasal Congestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Wave Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-008
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Nasal Congestion and Inflammations
MeSH Terms: conditions — Nasal Obstruction; Inflammation | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Ages 12-15 (Other): Pediatric subjects aged 12-15 years
  Interventions: Device: Acoustic Resonance (Sound) Therapy
- Ages 16-21 (Other): Pediatric subjects aged 16-21 years
  Interventions: Device: Acoustic Resonance (Sound) Therapy

INTERVENTIONS:
Device: Acoustic Resonance (Sound) Therapy — Sonu consists of an acoustic Vibrational Headband worn circumferentially at the level of the forehead; and a Smartphone App, paired to the Headband. The App determines acoustic resonant frequencies of the subject's nasal cavity (using the facial image) and delivers treatment through bone conduction transducers in the headband

SUMMARY:
To demonstrate the safety and effectiveness of Sonu for the treatment of pediatric patients with moderate to severe nasal congestion.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects between the ages of 12 to 21 years
* Present with symptoms of nasal congestion for 1 month or more prior to treatment
* Have a 24 hour reflective nasal congestion subscore of the TNSS of 2 or more on a 0 to 3 scale at the time of screening

Exclusion Criteria:

* Head, nasal or sinus surgery within 3 months
* Sinus infection diagnosed within the last month, or rhinitis medicamentosa
* Documented history of nasal polyposis or mass
* Pregnancy

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Serious adverse events | 2 weeks
  Safety
Reduction in nasal congestion subscore | 2 weeks
  Effectiveness

SECONDARY OUTCOMES:
Adverse events | 2 weeks
  Safety
Total Nasal Symptom Score (TNSS) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan Greene, MD, Principal Investigator — Crescendo MD
Locations (1):
- Crescendo MD, Portola Valley, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luong AU, Yong M, Hwang PH, Lin BY, Gopi P, Mohan V, Ma Y, Johnson J, Yen DM, DeMera RS, Bleier BS. Acoustic resonance therapy is safe and effective for the treatment of nasal congestion in rhinitis: A randomized sham-controlled trial. Int Forum Allergy Rhinol. 2024 May;14(5):919-927. doi: 10.1002/alr.23284. Epub 2023 Oct 9. PMID 37812532